CLINICAL TRIAL: NCT04700345
Title: Managing Non-acute Subdural Hematoma Using Liquid Materials：a Chinese Randomized Trial of MMA Treatment
Acronym: MAGIC-MT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Municipal Health Commission (Unknown); Shanghai Shen Kang Hospital Development Center (Other)
Responsible Party: Principal Investigator, Ying Mao, MD, PhD, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAGIC-MT
Record Dates: First submitted 2021-01-04; First posted 2021-01-07 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-08

CONDITIONS: Subdural Hematoma, Non-acute
MeSH Terms: conditions — Hematoma, Subdural | interventions — Trephining; Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Embolization (Experimental): Middle meningeal artery(MMA) embolization
  Interventions: Device: Onyx; Procedure: Burr-hole; Other: Medical Management
- No embolization (Active Comparator): Traditional treatment group
  Interventions: Procedure: Burr-hole; Other: Medical Management

INTERVENTIONS:
Device: Onyx — Embolization of the Middle Meningeal Artery using the liquid embolic material
  Arms: Embolization
Procedure: Burr-hole — Burr-hole drainage of subdural hematoma
Other: Medical Management — best medical management

SUMMARY:
MAGIC-MT study is multi-center, prospective, randomized (1:1) controlled trial designed to show that additional MMA embolization with Onyx in patients with non-acute symptomatic subdural hematoma(SDH) results in reduced hematoma recurrence in surgically treated patients/ reduced hematoma progression in conservatively managed patients.

DETAILED DESCRIPTION:
The objective of this study is to show that additional MMA embolization with Onyx in patients with non-acute symptomatic subdural hematoma(SDH) results in reduced hematoma recurrence in surgically treated patients/ reduced hematoma progression in conservatively managed patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic non-acute SDH with mass effect (i.e., chronic or subacute SDH)

   1. Mass effect refers to a shift in midline structure or deformation of local cerebral cortex due to SDH.
   2. Symptomatic defined as neurological symptoms, such as headache, short-term cognitive dysfunction, language disorder or aphasia, gait instability, decreased muscle strength, sensory disturbances, epileptic seizure, etc.
2. Age ≥18 years;
3. Pre-morbid mRS score 2;
4. Informed Consent Form (ICF) signed by patient or guardian.

Exclusion Criteria:

1. Radiographic imaging indicating massive cerebral infarction with corresponding symptoms;
2. Required craniotomy or craniotomy with small bone flap to remove SDH;
3. Emergency SDH removal/drainage;
4. Bilateral SDH with unknown origin of symptoms;
5. Anatomical variations that may affect the safety of MMA embolization (e.g., prominent middle MMA-ophthalmic artery anastomosis);
6. Intractable coagulation dysfunction or abnormal platelet count and function (pre-operative International Normalized Ratio [INR] > 1.5 and/or platelet count < 80109/L);
7. Contraindications to cerebral angiography, such as allergy to iodinated contrast agents, renal insufficiency (GFR < 30 ml/min), etc.;
8. Computed tomography (CT) or magnetic resonance imaging (MRI) showing intracranial space-occupying lesions;
9. Pregnancy or planning to become pregnant;
10. Serious or fatal coexisting disease that may prevent improvement of conditions or completion of follow-up;
11. Life expectancy < 1 year;
12. Recent operation unrelated to this study or investigators believe that they will be at higher risks if antiplatelet and/or anticoagulant drugs are discontinued;
13. Inability to complete follow-up as required by the protocol;
14. Patients participating in other clinical trials;
15. Prior surgery or interventional therapy on target SDH;
16. Inability to complete MMA embolization before trepanation and drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-06-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic SDH recurrence/ progression within 90 days post-procedure | 90 days
  SDH recurrence (>10 mm max. thickness) or receiving re-operation in patients who underwent surgery/ symptomatic SDH progression (>3 mm increase in max thickness or receiving surgical rescue in patients who did not undergo sugery) at 90 days
  "Symptomatic" is hereby defined as one or more of the following features which are attributed to the progression/recurrence: headache, short-term cognitive decline, speech difficulty or aphasia, gait impairment, focal weakness, sensory deficits, seizures

SECONDARY OUTCOMES:
Effectiveness | 1 year post-procedure
  Incidence of SDH recurrence/ progression at 1 year post-procedure
Effectiveness | day 0
  Rate of successful embolization of the target vessels (MMA trunk and branches) with ONYX base on DSA imaging
Effectiveness | 90 days post-procedure
  Change in hematoma thickness based on CT/MRI imaging at 90 days post-procedure
Effectiveness | 90 days post-procedure
  Changes in hematoma volume at 90 days post-procedure
Effectiveness | 90 days post-procedure
  Change in Midline shift based on CT/MRI imaging at 90 days post-procedure
Effectiveness | 90 days and 1 year post-procedure
  Change in the Modified Rankin Scale score (mRS) Grade 0 (no symptoms) to 6 (death) at 90 days and 1 year post-procedure
Effectiveness | 90 days and 1 year post-procedure
  Percentage of patients with favorable functional outcome defined as Modified Rankin Scale of 0 to 3 at 90 days and 1year post-procedure
Effectiveness | 90 days and 1 year post-procedure
  Percentage of patients with good functional outcome defined as Modified Rankin Scale of 0 to 2 at 90 days and 1 year post-procedure
Effectiveness | 90 days and 1 year post-procedure
  Quality of life assessed by (EuroQol) EQ-5D scale Grade 0 (worst health) to 100 (best health) at 90 days and 1 year post-procedure
Safety endpoint | 90 days
  Total patients with SAEs within 90 days post-procedure
Safety endpoint | 90 days
  Incidence of neurological death within 90 days post-procedure
Safety endpoint | 30 days
  Incidence of procedural serious complications within 30 days post-procedure:
  * symptomatic procedure-related intracranial hemorrhage
  * any procedure-related intracranial hemorrhage
  * any procedure-related neurological deficit
  * CNS infection caused by procedure
  * procedure-related artery dissection, vessel wall damage and vessel perforation
  * procedure-related ischemic event
  * retroperitoneal hematoma (femoral access)/wrist hematoma (radial access)
  * neuropathy at the puncture site
  * contrast agent allergy or encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Ying Mao, PhD, Principal Investigator — department of Neurosurgery, Huashan Hospital,Fudan University; Jian Min Liu, MD, Principal Investigator — Neurovascular Center, Trauma Center, Changhai Hospital, Naval Medical University
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu J, Ni W, Zuo Q, Yang H, Peng Y, Lin Z, Li Z, Wang J, Zhen Y, Luo J, Lin Y, Chen J, Hua X, Lu H, Zhong M, Liu M, Zhang J, Wang Y, Wan J, Li Y, Li T, Mao G, Zhao W, Gao L, Li C, Chen E, Cheng X, Zhang P, Wang Z, Chen L, Zhang Y, Tian B, Shen F, Lei Y, Wu Y, Li Y, Duan G, Xu L, Lv N, Yu J, Xu X, Du Z, Zhang H, Hu J, Li Z, Yuan Q, Zhou Y, Wu G, Zhang L, Gao C, Dai D, Wu X, Zhang Y, Jiang H, Zhao R, Su J, Xu Y, Ospel JM, Majoie CBLM, Goyal M, Li Q, Yang P, Gu Y, Mao Y; MAGIC-MT Investigators. Middle Meningeal Artery Embolization for Nonacute Subdural Hematoma. N Engl J Med. 2024 Nov 21;391(20):1901-1912. doi: 10.1056/NEJMoa2401201. PMID 39565989
- [Derived] Zuo Q, Ni W, Yang P, Gu Y, Yu Y, Yang H, Majoie CBLM, Goyal M, Liu J, Mao Y; MAGIC-MT investigators. Managing non-acute subdural hematoma using liquid materials: a Chinese randomized trial of middle meningeal artery treatment (MAGIC-MT)-protocol. Trials. 2023 Sep 14;24(1):586. doi: 10.1186/s13063-023-07608-2. PMID 37710274

DOCUMENTS (2):
  • Study Protocol (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT04700345/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT04700345/SAP_001.pdf